CLINICAL TRIAL: NCT01819415
Title: Omega-3 Supplementation and Vitreal VEGF Levels in Wet-AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Fonds de recherche en ophtalmologie de l'Université de Montréal (Other); Foundation Fighting Blindness (Other); Retina Foundation of Canada (Unknown); Insight Instruments (Unknown); Synergetics Inc (Unknown); Novartis (Industry)
Responsible Party: Principal Investigator, Flavio Rezende, Chief of Retina Service, Department of Ophthalmology, University of Montreal, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR-10059
Record Dates: First submitted 2013-03-24; First posted 2013-03-27 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Exudative Age Related Macular Degeneration
Keywords: wet AMD; Omega-3; VEGF; Lipidomics; DHA; EPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Naive (No Intervention): Patients starting on intravitreal anti-VEGF treatment, not receiving Omega-3 supplements. They serve as wet-AMD controls.
- Anti-VEGF plus AREDS-1 supplementation. (Active Comparator): Patients already receiving intravitreal anti-VEGF treatment assigned to take AREDS-1 plus Lutein supplementation formula.
  Interventions: Dietary Supplement: Anti-VEGF plus AREDS-1
- Anti-VEGF plus AREDS-2 (Experimental): Patients already receiving intravitreal anti-VEGF treatment assigned to take AREDS-2 supplementation formula, that includes Omega-3 metabolites (DHA and EPA).
  Interventions: Dietary Supplement: Anti-VEGF plus AREDS-2
- Control (No Intervention): Patients undergoing vitrectomy surgery for epiretinal membrane or macular hole had their vitreous samples to serve as controls.

INTERVENTIONS:
Dietary Supplement: Anti-VEGF plus AREDS-2 — Omega-3 metabolites supplementation
  Arms: Anti-VEGF plus AREDS-2
Dietary Supplement: Anti-VEGF plus AREDS-1 — Patients receiving intravitreal anti-VEGF and AREDS-1 supplementation plus Lutein, without Omega-3.
  Arms: Anti-VEGF plus AREDS-1 supplementation.

SUMMARY:
The purpose of this trial is to detect the influence of omega-3 supplements on vitreous levels of vascular endothelial growth factor (VEGF) in exudative age-related macular degeneration (AMD) in patients receiving intravitreal anti-VEGF treatment. Patients are randomized to receive either Age-Related Eye Disease Study 1(AREDS-1) supplements formula with the addition of Lutein or AREDS-2 supplementation that adds Omega-3 metabolites (DHA and EPA) to the formula. Our goal is to take a limited volume of vitreous sample from these patients previous to their regular anti-VEGF injection and perform a comprehensive cytokines and lipidomic profiling. We hypothesize, based on our previous basic science discovery of a potent anti-VEGF action of an Omega-3 metabolite (4-HDHA), that lipid metabolite composition and metobolite levels will significantly vary according to VEGF levels. Based on the results of this pioneering clinical study, our research team will proceed to evaluate the individual anti-angiogenic (vessel growth stopping) properties of the predominant Omega-3 metabolites found.

DETAILED DESCRIPTION:
The purpose of this trial is to detect the influence of omega-3 supplements on vitreous levels of vascular endothelial growth factor (VEGF) in exudative age-related macular degeneration (AMD) in patients receiving intravitreal anti-VEGF treatment. Patients are randomized to receive either Age-Related Eye Disease Study 1(AREDS-1) supplements formula with the addition of Lutein or AREDS-2 supplementation that adds Omega-3 metabolites (DHA and EPA) to the formula. Our goal is to take a limited volume of vitreous sample from these patients previous to their regular anti-VEGF injection and perform a comprehensive cytokines and lipidomic profiling. We hypothesize, based on our previous basic science discovery of a potent anti-VEGF action of an Omega-3 metabolite (4-HDHA), that lipid metabolite composition and metobolite levels will significantly vary according to VEGF levels.

ELIGIBILITY:
Inclusion Criteria:

* wet AMD eligible for intravitreal anti-VEGF treatment.
* Confirmed exudation on SD-OCT.

Exclusion Criteria:

* dry AMD.
* Disciform scar.
* Smokers.
* Morbid obesity.
* Patients undergoing other forms of treatment for wet AMD.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio A Rezende, MD, PhD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: February-August 2011 Location: Maisonneuve-Rosemont Hospital, University of Montreal, Quebec, Canada
Pre-assignment Details: At least 3 months of no other treatments for wet-AMD in groups 1 and 2 and no treatment at all for group 3.
Groups:
- Group 3 - Naive: Patients starting on intravitreal anti-VEGF treatment, not receiving Omega-3 supplements. They serve as wet-AMD controls.
- Group 2 - Anti-VEGF Plus AREDS-1 Supplementation.: Patients already receiving intravitreal anti-VEGF treatment assigned to take AREDS-1 plus Lutein supplementation formula.
- Group 1 - Anti-VEGF Plus AREDS-2: Patients already receiving intravitreal anti-VEGF treatment assigned to take AREDS-2 supplementation formula, that includes Omega-3 metabolites (DHA and EPA).
- Group 4 - Control: Patients undergoing vitrectomy surgery for epiretinal membrane or macular hole had their vitreous samples to serve as controls.
Period: Overall Study
Arm/Group | Group 3 - Naive | Group 2 - Anti-VEGF Plus AREDS-1 Supplementation. | Group 1 - Anti-VEGF Plus AREDS-2 | Group 4 - Control
Started | 10 | 10 | 10 | 10
Completed | 7 | 6 | 9 | 8
Not Completed | 3 | 4 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 3 - Naive | Group 2 - Anti-VEGF Plus AREDS-1 Supplementation. | Group 1 - Anti-VEGF Plus AREDS-2 | Group 4 - Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 83.38 (2.32) | 79.00 (1.98) | 79.6 (1.81) | 68.25 (3.56) | 77.56 (2.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 8 | 20
  Male | 7 | 6 | 5 | 2 | 20
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Vitreal VEGF Levels.
Time Frame: 1 day (At the time of vitreous biopsy)
Measure: Number; unit: pg/ml
Arm/Group | Group 3 - Naive | Group 2 - Anti-VEGF Plus AREDS-1 Supplementation. | Group 1 - Anti-VEGF Plus AREDS-2 | Group 4 - Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
pg/ml | 735.48 | 626.09 | 141.11 | 235.81

2. Primary Outcome: Lipidomics Profile
Time Frame: 1 day (At the time of vitreous biopsy)
Reporting Status: Not Posted

3. Secondary Outcome: Central Foveal Thickness
Description: Measured with spectral-domain optical coherence tomography.
Time Frame: During at least 12 months of follow-up after vitreous biopsy.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Group 3 - Naive | Group 2 - Anti-VEGF Plus AREDS-1 Supplementation. | Group 1 - Anti-VEGF Plus AREDS-2 | Group 4 - Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No